CLINICAL TRIAL: NCT05303766
Title: Comparing the Safety and Effectiveness of Radiofrequency Thermocoagulation on Genicular Nerve, Intraarticular Pulsed Radiofrequency With Steroid Injection in the Pain Management of Knee Osteoarthritis
Brief Title: Radiofrequency Ablation in the Pain Management of Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Mostafa Ali Osman, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Radiofrequency Ablation KOA
Record Dates: First submitted 2022-01-26; First posted 2022-03-31 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Radiofrequency Ablation; Steroids; Pulsed Radiofrequency Treatment

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RFT group (Experimental): The treatment of the patients in the radio frequency thermo-coagulation of the genicular nerves was conducted under the guidance of C-arm X-ray machine . The C-arm machine showed that the radiofrequency cannula needle was advanced percutaneously towards the periosteal areas connecting the shaft of the femur to bilateral epicondyles and the shaft of the tibia to the medial epicondyle while the lateral image showed that the depth of the needle insertion was about 50% of the diameter of the femur or tibia. The radiofrequency electrodes were connected and tested. These induced abnormal pain around the knee joint at 50 Hz and 0.1-0.3 V, but did not induce contraction of the muscles of the knee joint at 2 Hz and > 2.0 V. The location of the needle tip was confirmed by the C-arm, and 0.5 mL of 1% lidocaine was used for local anesthesia. The temperature of RFT was increased gradually to 70°C for 180 seconds.
  Interventions: Device: Radio-frequency ablation
- IAPRF group (Experimental): The puncture site was selected in the middle of the medial or lateral edge of the patella. After local anesthesia was administered with 0.5% lidocaine, the radiofrequency cannula needle was inserted slowly between the patella and femoral condyles. The needle was gradually inserted into the joint cavity, and then a small volume of saline was administered using a syringe. If any resistance was encountered, which indicated that the needle tip was located in a ligament or tendon, the surgeon readjusted the needle tip until the injection proceeded without any significant resistance. After entering the joint cavity, the C-arm x-ray is used confirm that the cannula needle was located in the middle of the joint space. Subsequently, sensory stimulation using 50 Hz/2 Hz was performed at > 2 V, to prevent inducing pain or muscle contraction. Then, an automatic PRF mode ≤ 45 V (≤ 42°C, 2 Hz, pulse width of 20 ms) was administered for 300 seconds.
  Interventions: Device: Pulsed Radio-frequency
- IAS group (Experimental): The puncture procedure was similar to that for the IAPRF group. After the cannula needle was inserted to the articular cavity, 1 mL compound betamethasone (2 mg betamethasone sodium phosphate and 5 mg betamethasone dipropionate) was injected. Then, the needle was withdrawn, and the puncture site was dressed aseptically.
  Interventions: Drug: Intra-articular steroids

INTERVENTIONS:
Device: Radio-frequency ablation — Radiofrequency thermocoagulation of the genicular nerves
  Other Names: Radiofrequency generator
  Arms: RFT group
Drug: Intra-articular steroids — Intra-articular steroids for Knee osteoarthritis
  Other Names: Betafos®
  Arms: IAS group
Device: Pulsed Radio-frequency — Intraarticular Pulsed Radiofrequency of the knee
  Other Names: Radiofrequency generator
  Arms: IAPRF group

SUMMARY:
The aim of this study is to assess the safety and efficacy of radio frequency thermo-coagulation on the genicular nerve (RFTGN) and intra-articular pulsed radio frequency (IAPRF) for Knee Osteoarthritis (KOA) to improve physical activity , range of joint movement , pain intensity and quality of life.

DETAILED DESCRIPTION:
After obtaining the consent from patients and being informed about the study and potential risks , all patients were randomly assigned to the RFTGN, IAPRF, and intraarticular steroid injection (IAS) groups. All procedures were performed under the guidance of C-arm X-ray machine. The observation indicators of this study were the numeric rating scale (NRS), Oxford knee scale (OKS), and perceived global effect (GPE). The time points for the assessment were 1-week, 1-month, 3-months, 6-months and 9-months after the treatment.

ELIGIBILITY:
* Inclusion Criteria:

  1. patients diagnosed with KOA based on the American College of Rheumatology criteria
  2. age 18-70 years
  3. grade 2 or 3 KOA based on the Kellgren-Lawrence classification
  4. patients who did not respond to conservative treatment (physiotherapy, oral NSAIDs, and/or intraarticular injections of hyaluronic acid and corticosteroid) for 3 months
  5. duration of knee pain ≥ 3 months
  6. numeric rating scale (NRS) ≥ 5 points within 24 h prior to admission.
* Exclusion Criteria:

  1. grade 1 or 4 KOA based on the Kellgren-Lawrence classification
  2. severe liver, kidney, cardiovascular, and respiratory disease
  3. abnormal blood coagulation
  4. skin infections in the puncture region
  5. patients who previously underwent knee arthroscopy, TKA, RFTGN, or IAPRF
  6. mental disorders or inability to complete the follow-up observational form
  7. patients with bilateral knee pain.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) | 9 months and after procedure
  Using the numerical rating score , a score from ( 0 to 10 ) for evaluation of pain intensity. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Oxford Knee Score | 9 months and after procedure
  Using oxford knee score for follow up of pain of knee osteoarthritis , a score from 0 to 48 . if the score is 0 to 19 this may indicate sever arthritis , and if it's from 40 to 48 it means satisfactory joint function . This scrore is based on a 12-question report about an individual's level of function, activities of daily living and how they have been affected by pain over the preceding four weeks.

SECONDARY OUTCOMES:
Duration of pain free periods | 9 months and after procedure
  Duration of pain free periods since the intervention has been done
Site of pain | 9 months and after procedure
  Patients undergo physical knee examination to determine the site of knee pain at right or left knee , medial or lateral joint line
Total consumption of analgesics ( e.g NSAIDS , weak opioids… ect ) | 9 months and after procedure
  Different analgesics used by the patients to alleviate the pain. The patient is asked about how frequent he/she uses an analgesic for pain relief.
Improvement of knee joint function | 9 months and after procedure
  Using The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) for evaluation of knee osteoarthritis. t is a self-administered questionnaire consisting of 24 items divided into 3 subscales: 1- Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright.
  2-Stiffness (2 items): after first waking and later in the day. 3- Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties.

CONTACTS AND LOCATIONS:
Overall Officials: Esraa M Osman, MBBCH, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD to be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting in March 2023
Access Criteria: Open access